CLINICAL TRIAL: NCT03786289
Title: Single Administration of Recombinant Human Serum Albumin/Erythropoietin Fusion Protein for Injection, Tolerance, Safety, Pharmacokinetics and Pharmacodynamic Clinical Trials of Increased Dosage
Brief Title: Study on Single Administration and Dose Increment of Recombinant Human Serum Albumin/Erythrocyte Fusion Protein for Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin SinoBiotech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1882-I
Record Dates: First submitted 2018-12-16; First posted 2018-12-26 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Healthy Subjects
Keywords: Recombinant human erythropoietin
MeSH Terms: interventions — Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant human serum albumin/erythropoietin fusion protein (Experimental): Recombinant human serum protein/erythropoietin fusion protein 150μg-1200μg single subcutaneous injection
  Interventions: Biological: Recombinant human serum albumin/erythropoietin fusion protein
- Recombinant human erythropoietin injection (CHO cells) (Active Comparator): Recombinant erythropoietin injection (CHO cells) 10000IU single subcutaneous injection
  Interventions: Biological: Recombinant erythropoietin injection (CHO cells)

INTERVENTIONS:
Biological: Recombinant human serum albumin/erythropoietin fusion protein — Recombinant human serum protein/erythropoietin fusion protein 150μg-1200μg single subcutaneous injection at Day1
  Arms: Recombinant human serum albumin/erythropoietin fusion protein
Biological: Recombinant erythropoietin injection (CHO cells) — Recombinant erythropoietin injection (CHO cells) 10000IU single subcutaneous injection at Day1
  Arms: Recombinant human erythropoietin injection (CHO cells)

SUMMARY:
The purpose of the study was to evaluate the safety of rHSA/EPO to healthy subjects and to investigate the pharmacokinetic characteristics of rHSA/EPO in healthy subjects, and to obtain preliminary pharmacokinetic parameters.

DETAILED DESCRIPTION:
This experiment was a single-center clinical study with randomized, open, positive drug control and single dose increment. The test group will be conducted in the order of incremental dose from 150μg to 1200μg 5 dose groups, with 1 positive control groups (EPIAO). After 7 days of administration, the researchers looked at the drug safety tolerance of the test to determine whether to proceed with the next higher dose group test.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) in the range of 19.0~26.0 (including critical value) (bmi= bw (kg)/ Height 2 (m2), male weight should be ≥50kg, female weight should be ≥45kg
* Understand and sign the informed consent form

Exclusion Criteria:

1. Persons with allergic physique or sensitive skin;
2. Any person with any skin disease;
3. have a history of drug or food allergies, especially for the active ingredients of this product or similar drugs, mammalian cells to The source of the drug, human serum albumin or other biological agents expressed in CHO allergy;
4. Pre-Test medical history, vital signs, physical examination, laboratory examination and other relevant examinations during the screening period, Abnormal and clinically significant person;
5. Previous intentional cerebral vessels, liver, kidneys, lungs, digestive tract, nerves, autoimmune, metabolic and skeletal muscle system, hematopoietic system and other diseases of history;
6. Having a fertility plan within 2 weeks of screening and within 6 months of the end of the trial and not having to take it during the trial period

   (a) Effective non-drug contraceptive measures;
7. Within 14 days prior to screening or within 5 half-life of the drug (whichever is the oldest of the two) there has been any Prescription drugs, over-the-counter drugs, Chinese herbal medicine, health care products medicine history;
8. Hemoglobin ≤130 g/L or ≥150/g (male), hemoglobin ≤115 g/L or ≥133 g/L (female version number: 1.2 Version date: September 30, 2018 26 sexual);
9. The percentage of erythrocyte red blood cells ≥ 3%;
10. ferritin <200 ng/ml (male), ferritin <80 ng/ml (female);
11. The use of drugs known to have damage to an organ during the first 3 months of screening;
12. A person who has received a blood transfusion or rhEPO treatment;
13. Clinically determined to be vitamin B12 or folic acid deficiency;
14. Have a history of dizziness and needle sickness;
15. A clinical trial person who has participated in other drugs within the first 3 months of screening;
16. Those who had lost blood or blood ≥200ml during the first 8 weeks of screening;
17. Women during pregnancy and lactation;
18. The researchers did not consider it appropriate to enter the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Day1-Day29
  Incidence of adverse events, adverse reactions and serious adverse events after single administration

SECONDARY OUTCOMES:
Concentration of recombinant human serum albumin/erythrocyte fusion protein in serum | Day1-Day29
  Rhsa/epo: Before administration, after administration 1h,2h,6h,12h,24h(2nd day), 36h(2nd day), 48h(3rd day), 72h(4th day), 96h(5th day), 120h( Day 6th), 168h(day 8th), 336h(Day 15th), 504h(22nd days) and 672h (29th days) Blood collection measures drug concentrations.
Concentration of recombinant human erythropoietin injection (Cho cell) in serum | Day1-Day29
  Recombinant human erythropoietin injection (Cho cells): Before and after administration, 1h,2h,6h,9h,12h,18h,24h(2nd day), 36h(2nd day), 48h(3rd day), 72h(4th day), 96h(5th day), 120h( Day 6th), 168h(day 8th), 336h(Day 15th), 504h(22nd days) and 672h (29th days) Blood collection measures drug concentrations.
Erythrocyte count,before and after administration | Day1-Day29
  Rhsa/epo: Before administration, after administration 1h,2h,6h,12h,24h(2nd day), 36h(2nd day), 48h(3rd day), 72h(4th day), 96h(5th day), 120h( Day 6th), 168h(day 8th), 336h(Day 15th), 504h(22nd days) and 672h (29th days) Blood collection measures red blood cell counts.
  Recombinant human erythropoietin injection (Cho cells): Before and after administration, 1h,2h,6h,9h,12h,18h,24h(2nd day), 36h(2nd day), 48h(3rd day), 72h(4th day), 96h(5th day), 120h( Day 6th), 168h(day 8th), 336h(Day 15th), 504h(22nd days) and 672h (29th days) Blood collection measures red blood cell counts.
hemoglobin,before and after administration | Day1-Day29
  Rhsa/epo: Before administration, after administration 1h,2h,6h,12h,24h(2nd day), 36h(2nd day), 48h(3rd day), 72h(4th day), 96h(5th day), 120h( Day 6th), 168h(day 8th), 336h(Day 15th), 504h(22nd days) and 672h (29th days) Blood collection measures hemoglobin concentrations.
  Recombinant human erythropoietin injection (Cho cells): Before and after administration, 1h,2h,6h,9h,12h,18h,24h(2nd day), 36h(2nd day), 48h(3rd day), 72h(4th day), 96h(5th day), 120h( Day 6th), 168h(day 8th), 336h(Day 15th), 504h(22nd days) and 672h (29th days) Blood collection measures hemoglobin concentrations.
the percentage of erythrocyte red blood cells,before and after administration | Day1-Day29
  Rhsa/epo: Before administration, after administration 1h,2h,6h,12h,24h(2nd day), 36h(2nd day), 48h(3rd day), 72h(4th day), 96h(5th day), 120h( Day 6th), 168h(day 8th), 336h(Day 15th), 504h(22nd days) and 672h (29th days) Blood collection measures the percentage of erythrocyte red blood cells.
  Recombinant human erythropoietin injection (Cho cells): Before and after administration, 1h,2h,6h,9h,12h,18h,24h(2nd day), 36h(2nd day), 48h(3rd day), 72h(4th day), 96h(5th day), 120h( Day 6th), 168h(day 8th), 336h(Day 15th), 504h(22nd days) and 672h (29th days) Blood collection measures the percentage of erythrocyte red blood cells.
erythrocyte ratio (HCT) before and after administration | Day1-Day29
  Rhsa/epo: Before administration, after administration 1h,2h,6h,12h,24h(2nd day), 36h(2nd day), 48h(3rd day), 72h(4th day), 96h(5th day), 120h( Day 6th), 168h(day 8th), 336h(Day 15th), 504h(22nd days) and 672h (29th days) Blood collection measures blood cell accumulations.
  Recombinant human erythropoietin injection (Cho cells): Before and after administration, 1h,2h,6h,9h,12h,18h,24h(2nd day), 36h(2nd day), 48h(3rd day), 72h(4th day), 96h(5th day), 120h( Day 6th), 168h(day 8th), 336h(Day 15th), 504h(22nd days) and 672h (29th days) Blood collection measures blood cell accumulations.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing you 'an hospital affiliated to capital medical university, Beijing, Beijing Municipality, China